CLINICAL TRIAL: NCT05472987
Title: Robotic Versus Open Ventral Hernia Repair: A Randomized Controlled Trial
Brief Title: Robotic Versus Open Ventral Hernia Repair
Acronym: ROVHR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lucas Beffa (Other)
Responsible Party: Sponsor-Investigator, Lucas Beffa, Assistant Professor of Surgery, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22-591
Record Dates: First submitted 2022-07-20; First posted 2022-07-25 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Ventral Hernia
Keywords: Robotic; Hernia; Ventral hernia; Open hernia; Mesh
MeSH Terms: conditions — Hernia, Ventral; Hernia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to the intervention. The primary outcome will be determined by a surgeon other than the operating surgeon who is blinded to the intervention. Patients will also receive the same dressings over their wounds and an abdominal binder will be placed over the abdomen in attempts to limit the unblinding of the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open Ventral Hernia Repair (Active Comparator): These patients will undergo open retromuscular ventral hernia repairs
  Interventions: Procedure: Ventral Hernia Repair
- Robotic Ventral Hernia Repair (Active Comparator): These patients will undergo robotic retromuscular ventral hernia repairs.
  Interventions: Procedure: Ventral Hernia Repair

INTERVENTIONS:
Procedure: Ventral Hernia Repair — Patients will undergo retromuscular ventral hernia repair

SUMMARY:
This is a randomized trial comparing open retromuscular ventral hernia repair to robotic retromuscular ventral hernia repair.

DETAILED DESCRIPTION:
This is a randomized trial comparing open retromuscular ventral hernia repair to robotic retromuscular ventral hernia repair. This is a superiority trial with a primary outcome of length of stay in the hospital, theorizing that robotic retromuscular ventral hernia repairs are superior to open ventral hernia repairs by reducing length of stay by 24 hours. Patients will be blinded to the intervention, groups will be in parallel, and the primary outcome (when the patient is discharged) will be determined by a blinded assessor.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* 7 cm to 15 cm wide hernia midline defects
* BMI less than or equal to 45
* Patient deemed both an open and robotic candidate by operating surgeon

Exclusion Criteria:

* 17 years old or younger
* prisoners
* pregnant patients
* Emergent patients
* BMI greater than 45
* Hernia defects less than 7 cm or greater than 15 cm in width

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Length of Stay | 30 days
  Time in the hospital after the surgery

SECONDARY OUTCOMES:
Post-operative wound complications | 30 day and one year
  any abnormal wound healing
Other post operative complications | 30 days
  Heart attacks, acute kidney injury, admissions to ICU, respiratory failure
Readmission rate | 30 days
  Readmission to the hospital within 30 days of the surgery
Opioid consumption | 30 days and one year
  Opioid prescribed and consumed
Acute pain scores | 5 days after surgery
  Numeric Rating Scale-11 pain scores daily, 0-10 with 0 being no pain and 10 being the worst pain for first five days after surgery
Hernia Related Specific Quality of Life Score | 30 days and one year
  Score of 0-100 with lower scores indicating worse quality of life
Direct cost | 30 days
  Cost to the hospital
Hernia recurrence | 30 days and one year
  Hernia recurrence
Quality of life scores using European Hernia Society (EuraHS) scale | 30 day and one year
  EuraHS is a hernia specific quality of life scale with three domains: pain, restrictions of activity, and cosmesis. 0-30 with higher scores indicating a worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Lucas Beffa, MD, Principal Investigator — The Cleveland Clinic
Locations (4):
- United States (4):
  - University of Florida Health, Gainesville, Florida
  - Cleveland Clinic, Cleveland, Ohio
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - University of Tennessee Medical Center, Knoxville, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carvalho AC, Woo KP, Ellis RC, Tu C, Miller BT, Prabhu AS, Rosen MJ, Krpata DM, Petro CC, Beffa LR. Robotic versus open ventral hernia repair (ROVHR): a randomized controlled trial protocol. Hernia. 2025 Mar 4;29(1):109. doi: 10.1007/s10029-025-03299-7. PMID 40035894